CLINICAL TRIAL: NCT07322692
Title: The Effect of Nurse-Led PRECEDE-PROCEED Model-Based Risk Management Program on Reducing Musculoskeletal Symptoms in Primary School Children
Brief Title: Effect Nurse-Led PRECEDE-PROCEED Model Based Risk Management Program on Reducing Musculoskeletal Symptoms in Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Makbule Senel, Research Assistans, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: İUC-FNFN-MS-01
Record Dates: First submitted 2025-10-01; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Primary School Children; Musculoskeletal Symptom
Keywords: musculoskeletal symptom; primary school children

STUDY DESIGN:
Intervention Model Description: This study aims to determine the effect of the nurse-led PRECEDE-PROCEED model-based ergonomic risk management education program on reducing musculoskeletal symptoms in primary school children.
Who Masked: Participant
Masking Description: Participants in the study will not know whether they are in the experimental or control group. This information will remain confidential with the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will be given training on ergonomic risk factors.
  Interventions: Other: ergonomic risk management awareness training
- control grup (No Intervention): No attempt was made to initiate the training process

INTERVENTIONS:
Other: ergonomic risk management awareness training — For 4 weeks, the experimental group will be trained on ergonomic risk factors (moving in appropriate posture, using ergonomic desks and chairs, carrying a backpack of appropriate weight according to body mass index (BMI), etc.).
  Arms: Experimental group

SUMMARY:
The Effect of a Nurse-Led Ergonomic Risk Management Program Based on the PRECEDE-PROCEED Model on Reducing Musculoskeletal Symptoms in Primary School Children

DETAILED DESCRIPTION:
Primary school children spend a large portion of their school hours sitting at their desks (Chen 2021, Van Delden 2020). Students are associated with musculoskeletal pain and discomfort due to prolonged sitting (Guelfi 2019). Common causes of these musculoskeletal system (MSS) problems include carrying inappropriately heavy backpacks, sitting for extended periods in the classroom, long class hours, standardized desks and seats, excessive homework, and prolonged use of phones, tablets, and computers outside of homework. These factors contribute to MSS problems in children, particularly musculoskeletal pain and posture disorders. It is known that the prevalence of posture disorders in school children is increasing (Kinaci 2018). 55.5% of students reported having to lean over their desks while writing at school, and 58.1% reported discomfort due to the weight of their school bags (Yılmaz 2018). Because school-aged children are in the developmental stage of MSD and body posture is being shaped, if proper ergonomic adjustments and behavioral development interventions are not implemented during this period, significant health problems can occur in later years (Contardo 2016). Therefore, interest in school ergonomic intervention programs and their effects on MSD is increasing globally (Sellschop 2015). There is an urgent need for ergonomics-specific and behavior-based school programs (Ayed 2019). Research suggests that school nurses should be involved in these school health programs. To prevent MSD problems, they should collaborate with teachers to organize educational programs on posture training, weight-bearing methods, and the importance of exercise. They should also implement ergonomic adjustments in the classroom and regularly reiterate these recommendations with school administrators and guidance counselors (Yılmaz 2018). Therefore, this study aims to determine the effectiveness of a nurse-led ergonomic risk management education program based on the PRECEDE-PROCEED model on reducing MSD symptoms in primary school children.

ELIGIBILITY:
Inclusion Criteria:

* Being a student,
* Being in the 3rd or 4th grade,
* Volunteering to participate in the research,
* Volunteering with parental consent,
* No musculoskeletal problems,
* No physical disabilities that would prevent exercise,

Exclusion Criteria:

* Those diagnosed with a chronic disease
* Those with musculoskeletal problems
* Those with physical disabilities that may prevent them from exercising
* Those who volunteer but do not have parental permission
* Those who have parental permission but do not volunteer

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Evaluation | The 4th week
  It evaluates effort, repetition frequency, and duration of work at the upper arm, lower arm, wrist, neck, and trunk. Each site is assigned an Ergonomic Risk Score (ERP) from 1 to 4, with ERP 1 indicating acceptable risk, ERP 2 indicating risk requiring further investigation, ERP 3 indicating serious risk requiring immediate intervention and remediation, and ERP 4 indicating highest risk requiring immediate change.
Musculoskeletal Disorders Evaluation | The 4th week
  The survey assesses frequency, severity, and work-relatedness, and calculates a total discomfort score. Frequency is scored as "Never" = 0; 1-2 times a week = 1.5; 3-4 times a week = 3.5; Once a day = 5; Several times a day = 10; severity is scored as "little" = 1, moderate = 2, and severe = 3; and work-relatedness is scored as "little" = 1, moderate = 2, and severe = 3. The total discomfort score frequency x severity x work relevance of discomfort).

SECONDARY OUTCOMES:
Upper Extremity Evaluation | The 12th week
  It evaluates effort, repetition frequency, and duration of work at the upper arm, lower arm, wrist, neck, and trunk. Each site is assigned an Ergonomic Risk Score (ERP) from 1 to 4, with ERP 1 indicating acceptable risk, ERP 2 indicating risk requiring further investigation, ERP 3 indicating serious risk requiring immediate intervention and remediation, and ERP 4 indicating highest risk requiring immediate change.
Musculoskeletal Disorders Evaluation | The 12th week
  The survey assesses frequency, severity, and work-relatedness, and calculates a total discomfort score. Frequency is scored as "Never" = 0; 1-2 times a week = 1.5; 3-4 times a week = 3.5; Once a day = 5; Several times a day = 10; severity is scored as "little" = 1, moderate = 2, and severe = 3; and work-relatedness is scored as "little" = 1, moderate = 2, and severe = 3. The total discomfort score frequency x severity x work relevance of discomfort).

CONTACTS AND LOCATIONS:
Locations (1):
- Makbule Şenel, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2022- 2025
Access Criteria: 2025